CLINICAL TRIAL: NCT04500080
Title: Feasibility and Safety of Physical Exercise Program in Men With Prostate Cancer Receiving Androgen Deprivation Therapy and Radiotherapy
Brief Title: Feasibility and Safety of Physical Exercise in Men With Prostate Cancer
Acronym: PCa_Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Fondazione Manodori di Reggio Emilia (Unknown); University of Modena and Reggio Emilia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 520/2020/SPER/IRCCSRE
Record Dates: First submitted 2020-08-01; First posted 2020-08-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Androgen Deprivation Therapy; Radiotherapy
Keywords: Exercise; Feasibility; Safety
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PE intervention (Experimental): Aerobic, resistance, and neuromotor exercise
  Interventions: Behavioral: PE Intervention

INTERVENTIONS:
Behavioral: PE Intervention — Each single exercise session will last for one hour and will consist of a combination of the following elements:
  * Aerobic Exercise (AE): 20-30 minutes at moderate-high intensity, from 60 to 80% of the maximum heart rate (% HRmax).
  * Resistance Exercise (RE): 30 minutes of strength activity of the major muscle groups.
  * Neuromotor Exercise (NE): will be integrated with strength exercises and will consist of jumping, balance and coordination activities

SUMMARY:
Prostate cancer (PCa) is among the most widespread in the male population and represents 19% of all cancers diagnosed from the age of fifty, in Italy. Androgen deprivation therapy (ADT) and Radiotherapy (RT) are used for increase survival. However, both therapies are associated with significant side effects, such as fatigue, loss of muscle mass and strength, cognitive decline that together lead to an increase risk of accidental falls and fractures.

Guidelines for cancer survivors recommend Physical Exercise (PE) as a strategy to reduce several side effects of therapies. However, most people living with cancer do not meet current exercise recommendations.

Indeed, an effective PE program requires the application of long-term, moderate to high intensity activity. Thus it may be difficult to implement this type of recommendation in patient with PCa.

Therefore, this study aims to develop an experimental PE intervention testing their feasibility and safety and the patients' satisfaction, aimed at improving the health conditions of the patients with PCa receiving ADT and RT. Furthermore, long-term falls and fracture events will be monitored.

DETAILED DESCRIPTION:
The non-randomized feasibility and pilot study aims to evaluate the feasibility and safety of a structured, multicomponent, supervised and unsupervised exercise program.

Secondary outcome will be evaluate the change in the health condition, in particular muscle strength, cognitive function, fatigue, balance, anxiety and depression level, and quality of life.

The PE program will be conducted at the "Virgilio Camparada" Municipal Athletic Track in the city of Reggio Emilia (IT). Patients will be participate in a supervised exercise program with three sessions per week, for eight weeks. Subsequently, the intervention will continue further for four weeks maintaining one supervised session and two unsupervised sessions a week. Finally, sessions will be performed without supervision for further eight weeks. The overall duration of the intervention will be twenty weeks. In addition, an evaluation will be performed at one year from baseline to monitor long-term fall and fracture events.

At baseline will be the following assessment:

- clinical and anthropometric data and the Six Minute Walking Test (6MWT) to determine the intensity of aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of PCa;
* Undergo ADT and RT during the study period;
* At least 18 years old;
* Willing and able to give written informed consent;
* Able to read and understand Italian Language;

Exclusion Criteria:

* Musculoskeletal, cardiovascular, neurological or psychiatric disorders that contraindicate participation in an exercise program.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment rate | At baseline (T0)
  Percentage ratio between patients included in the study and number of participants screened for recruitment.
Feasibility - Adherence rate to the exercise program | Throughout the 20 week study period
  Determine the percentage of patients adhering to the program and the weekly exercise sessions.
Feasibility - Dropout rate | Throughout the 20 week study period
  Percentage of patients that withdraw from the study and the reason to withdraw
Feasibility - Safety/Adverse events | Throughout the 20 week study period
  Any adverse events, related or not related to the exercise program, will be documented
Feasibility - Compliance and patients' experience | Following the study conclusion at 20 weeks.
  Determined by qualitative evaluation, using interviews, to assess experiences, accessibility and acceptability of the exercise intervention.

SECONDARY OUTCOMES:
Change of muscular strength assessment | At baseline and 20 weeks.
  Lower body muscle strength will be determined with the 10-repetitions maximum test.
Change of cognitive status assessment | At baseline and 20 weeks.
  Cognitive status will be assess using the Mini Mental State Examination (MMSE), a 30-point questionnaire italian version. A score of 24 or more (out of 30) indicates a normal cognition.
Change of fatigue assessment | At baseline and 20 weeks.
  Fatigue will be measured using the Fatigue Severity Scale (FSS). FSS is a 9-item questionnaire on how fatigue interferes activities and rates its severity. The item are scored on a 7 point scale with 1 = strongly disagree and 7 = strongly agree. The minimum score = 9, maximum score = 63. Higher score means greater fatigue severity.
Change of fall risk assessment | At baseline and 20 weeks.
  Fall risk will be assessed using the Tinetti Performance Oriented Mobility Assessment (POMA). The Tinetti POMA is a clinical test used to measure balance and gait abilities. The balance section (POMA-B) consists of 9 items while the gait section (POMA-G) consists of 8 items.Each of these items has answer choices that are weighted on an ordinal scale from 0 to 1 or 2. "0" indicates the highest level of impairment and "2" the individuals independence. The maximum possible total score for POMA-T is 28, for POMA-B is 16, and for POMA-G is 12.
Change of anxiety and depression level | At baseline and 20 weeks.
  Depression and anxiety level will be measured using the Hospital Anxiety and Depression Scale (HADS). The HADS is a fourteen item scale, seven relate to anxiety and seven relate to depression. The total score goes from 0-21. Higher total scores indicate greater levels of depression.
Change of quality of life assessment | At baseline and 20 weeks.
  Quality of life will be measured by a Short form-12 questionnaire (SF-12). The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Higher scores indicate a better physical and mental health.
Falls and fractures. | Throughout the 20 week study period and at one year of follow-up.
  Registration of number of falls and fractures events through patient interview.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Costi, Ph.D., Principal Investigator — Azienda Unità Sanitaria Locale-IRCCS di Reggio Emilia
Locations (1):
- Azienda USL-IRCCS di Reggio Emilia, Reggio Emilia, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Winters-Stone KM, Moe E, Graff JN, Dieckmann NF, Stoyles S, Borsch C, Alumkal JJ, Amling CL, Beer TM. Falls and Frailty in Prostate Cancer Survivors: Current, Past, and Never Users of Androgen Deprivation Therapy. J Am Geriatr Soc. 2017 Jul;65(7):1414-1419. doi: 10.1111/jgs.14795. Epub 2017 Mar 6. PMID 28263373
- [Result] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Result] Feng LR, Espina A, Saligan LN. Association of Fatigue Intensification with Cognitive Impairment during Radiation Therapy for Prostate Cancer. Oncology. 2018;94(6):363-372. doi: 10.1159/000487081. Epub 2018 Mar 7. PMID 29514170
- [Result] Gardner JR, Livingston PM, Fraser SF. Effects of exercise on treatment-related adverse effects for patients with prostate cancer receiving androgen-deprivation therapy: a systematic review. J Clin Oncol. 2014 Feb 1;32(4):335-46. doi: 10.1200/JCO.2013.49.5523. Epub 2013 Dec 16. PMID 24344218
- [Result] Bourke L, Smith D, Steed L, Hooper R, Carter A, Catto J, Albertsen PC, Tombal B, Payne HA, Rosario DJ. Exercise for Men with Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Apr;69(4):693-703. doi: 10.1016/j.eururo.2015.10.047. Epub 2015 Nov 26. PMID 26632144
- [Derived] Bressi B, Iotti C, Cagliari M, Cavuto S, Fugazzaro S, Costi S. Feasibility and safety of physical exercise in men with prostate cancer receiving androgen deprivation therapy and radiotherapy: a study protocol. BMJ Open. 2022 Mar 15;12(3):e048854. doi: 10.1136/bmjopen-2021-048854. PMID 35292485